CLINICAL TRIAL: NCT00860587
Title: Risk Factors for Colonization and Infection With Antibiotic Resistant Bacteria Among Patients With Severe Intraabdominal Infections (IAI). An Open Observational Study
Brief Title: Antibiotic Resistant Bacteria Among Patients With Severe Intraabdominal Infections
Acronym: Bakki
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Linkoeping (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Professor Håkan Hanberger, Division of Infectious Diseases, University Hospital, SE-581 85 Linköping
Other Study IDs: Bakki
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2009-03

CONDITIONS: Complicated Intra-Abdominal Infections
Keywords: Antibiotic resistance; Antibiotic treatment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objectives of the study were:

1. To study risk factors for colonization and infection with antibiotic resistant bacteria among patients with severe IAI before and after antibiotic treatment and surgical intervention.
2. To study species changes in the rectal flora among patients with severe IAI before and after antibiotic treatment and surgical intervention.
3. To review guidelines for antibiotic use in participating units.
4. To evaluate surgical antibiotic prophylaxis and treatment in relation to risk for colonization and infection with antibiotic resistant bacteria among patients with severe IAI
5. To use the results from the study in the process of a more appropriate use of antibiotics in participating units and care of patients with severe IAI.
6. To study the dynamics of extended-spectrum beta-lactamase producing and wild-type Enterobacteriaceae in patients with suspected severe intra abdominal infections before, during and after antibiotic treatment.

DETAILED DESCRIPTION:
In order to evaluate if standard empirical treatment was adequate in relation to resistance pattern among most prevalent species at admission we need another 70 patients to be included with at least data and cultures from admission.

ELIGIBILITY:
Inclusion Criteria:

* Patients with evidence of intra-abdominal infections that require surgical intervention will be eligible.
* In addition will patients with intra-abdominal abscess confirmed with CT/ultrasound be eligible, but not treated with surgical intervention if estimated to require at least 5 days antibiotic treatment, with a severity needing initial intravenous administration of antibiotics.

Exclusion Criteria:

* Age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with evidence of severe intra-abdominal infections.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2006-02; Primary Completion 2009-10 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Primary End points for detection of AB-R Colonising index: (a) Proportion of patients colonised with AB-R strains per bacteria species.(b)Proportion of colonising cultures containing AB-R strains per bacteria species. | 48 hours - 2 weeks after end of antibiotic treatment

SECONDARY OUTCOMES:
Proportion of patients with SSI other postoperative infections caused by AB-R strains, per infection type and per bacteria species. | 48 hours - 2 weeks after end of antibiotic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Håkan SI Hanberger, Professor, Principal Investigator — Division of Infectious Diseases, University Hospital, Linköping